CLINICAL TRIAL: NCT02808338
Title: Servo-Ventilation In-lab Polysomnography (PSG) Evaluation
Brief Title: Servo-Ventilation In-lab PSG Evaluation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philips Respironics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ST-1517-ALE-MS
Record Dates: First submitted 2016-06-07; First posted 2016-06-21 (Estimated); Results first posted 2019-03-19 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2019-02

CONDITIONS: Sleep Apnea Syndromes
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (4):
- Philips BiPAP AutoSV Advanced System One (Active Comparator): The Bi-Level Positive Airway Pressure system will be used and will be configured with these settings.
  P max: 30 EPAP min: 4 EPAPmax: 15 Pressure Support (PS) min: 0 Pressure Support (PS) max: 15 BiFlex: 2 Rate: Auto
  Interventions: Device: Philips BiPAP AutoSV Advanced System One
- Modified Philips BiPAP ASV (Experimental): The modified Philips BiPAP ASV will be configured with these settings P max: 30 EPAP min: 4 EPAPmax: 15 PS min: 0 PS max: 15 BiFlex: 2 Rate: Auto
  Interventions: Device: Modified Philips BiPAP ASV
- ResMed S7 VPAP Adapt (Active Comparator): This is an FDA approved device and the following settings will be administered:
  End-expiratory Pressure (EEP): 4 PSmin: 3 PSMax: 16
  Interventions: Device: ResMed S7 VPAP Adapt
- ResMed S9 VPAP Adapt (Active Comparator): This is an FDA approved device and the following settings will be administered:
  EPAP min: 4 EPAPmax: 15 PS min: 0 PS max: 20 Max Ramp: Off
  Interventions: Device: ResMed S9 VPAP Adapt

INTERVENTIONS:
Device: Philips BiPAP AutoSV Advanced System One — Auto SV Auto Servo Ventilation is a mode of positive airway pressure used to treat obstructive and complex central sleep apnea. This devices is FDA approved and will be set according to a predetermined setting.
  Arms: Philips BiPAP AutoSV Advanced System One
Device: Modified Philips BiPAP ASV — This Modified BiPAP ASV will be set to a predetermined setting. This is the investigational device.
  Arms: Modified Philips BiPAP ASV
Device: ResMed S7 VPAP Adapt — This device is FDA approved and will be set to predetermined setting.
  Arms: ResMed S7 VPAP Adapt
Device: ResMed S9 VPAP Adapt — This device is FDA approved and will be set to predetermined setting.
  Arms: ResMed S9 VPAP Adapt

SUMMARY:
Continuous Positive Airway Pressure (CPAP) is the most effective treatment for the Obstructive Sleep Apnea-Hypopnea Syndrome (OSAHS). CPAP stabilizes the airway and prevents instability and collapse. With a stable and patent airway, breathing continues in a normal manner, gas exchange is improved, and there is no disruption of sleep related to disturbed breathing.

Auto Servo Ventilation (Auto SV) is a mode of positive airway pressure used to treat obstructive and complex central sleep apnea. The main features of the Auto SV mode include:

* Normalization of ventilation by automatically adjusting Inspiratory Positive Airway Pressure (IPAP) pressure to achieve a target ventilation. IPAP is increased or decreased to help stabilize the ventilation.
* Provision of timed, back-up breaths during central apneas. The optimal back-up rate is automatically determined by the device based on the patient's breathing.
* Automatic control of Expiratory Positive Airway Pressure (EPAP) to treat obstructive events.

Several manufacturers produce these types of devices. The algorithms used to determine the IPAP, EPAP and minimum respiratory rate are different. The largest number of these devices currently in use are the BiPAP AutoSV Advanced System One (Philips Respironics, Murrysville PA) and the Variable positive airway pressure (VPAP) Adapt (ResMed Corp., San Diego CA).

DETAILED DESCRIPTION:
This study is to better understand the performance and features of the BiPAP autoSV Advanced System One. Philips Respironics will evaluate the PolySomnoGraphy (PSG) and Encore data from each night. The aim of the study is to characterize the acute outcomes of treatment provided by the device and evaluate any modifications made to the Philips Respironics device's algorithm

The participants for this study will be experienced in having used servo ventilation therapy at their home because it is only such patients who are already using servo ventilation as part of routine clinical care that are eligible for participation.

Participants will receive four (4) randomized PSG's during which they will receive treatment from the following devices in a randomized manner:

* FDA released Philips BiPAP AutoSV Advanced System One
* A Modified Philips BiPAP ASV
* FDA released ResMed S7 VPAP Adapt
* FDA released ResMed S9 VPAP Adapt

The participants sought for this effort will be previously prescribed a servo-ventilation device as part of routine clinical care.

Baseline with PSG

* Informed Consent
* Inclusion/Exclusion Criteria Review
* Demographics
* Anthropometric Measurements
* PAP Prescription information (if available; from Device or from Medical records). This is the pressure settings of the device that was prescribed by the patient's clinical sleep medicine provider.
* Medical History and physical examination
* Sleep History- Including that past 30 day detailed report
* Diagnostic PSG history (copies of sleep studies that were performed as part of routine clinical care in the past that qualified the patient for the servo-ventilation device)
* Current Medications
* Vital Signs (at beginning of PSG night)
* Research Trial PSG- Randomized to a device Procedures for Each PSG after Baseline
* Current Medications
* Vital Signs (at beginning of PSG night)
* Research Trial PSG- Randomized to one of the four devices (4 research PSGs will be performed for each subject).

  30 day Take Home with Modified Philips BiPAP ASV device

After the last PSG participants will be sent home on Modified Philips Auto Servo Ventilation (ASV) study device. A wireless modem with oxygen saturation level (SPO2) connection will be connected to the Modified Philips ASV study device. The wireless modem with SPO2 connection is for device data collection/transmission purposes only that monitors the usage and performance of the device in the home-setting.

* The device setting should be set to the following:

  * P max: 30
  * EPAP min: 4
  * Expiratory Positive Airway Pressure maximum (EPAPmax):15
  * Pressure Support Minimum (PS min): 0
  * Pressure Support Maximum (PS max): 15
  * BiFlex (Bi-Level Flex): 2
  * Rate: Auto

After 30 day Take Home Participants Will

* Return to the Sleep Lab
* Complete the end of study questionnaire
* Return all of the study equipment

Additional Take Home with the Modified Philips BiPAP ASV device:

* Participants may be asked to use the Modified Philips ASV study device for an additional 30 days if more data is needed for analysis. Participants will complete the same end of day questionnaire noted above.

After trial completion:

* When the Participant is done with the trial they will go back to using their own prescribed device.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide consent
* Age ≥ 21
* Currently prescribed servo ventilation therapy at home
* At least two weeks of recent adherence and efficacy data from PAP device demonstrating adequate use of therapy (at least 4 hours of use per night and use on at least 9 of 14 nights)
* Current device compliance report demonstrating residual Apnea-Hypopnea Index (AHI) of 5 or more

Exclusion Criteria:

* Participants who are acutely ill, medically complicated or who are medically unstable
* Participants in whom PAP therapy is otherwise medically contraindicated
* Participants who are claustrophobic
* Symptomatic ("Symptomatic" defined as hospitalized for heart failure or a change in cardiac medications, within the last two months) chronic heart failure (NYHA 2-4) and reduced LVEF≤45%, AND moderate to severe predominant central sleep apnea
* Participants with previously diagnosed respiratory failure or respiratory insufficiency and who are known to have elevated arterial carbon dioxide levels while awake (PaCO2 ≥ 55mmHg).
* Participants requiring any kind of oxygen therapy
* Participants who have had surgery of the upper airway, nose, sinus, eyes, or middle ear within the previous 90 days
* Participants with untreated, non-OSA sleep disorders, including but not limited to; insomnia, periodic limb movement syndrome, or restless legs syndrome (PLMI > 10).

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2015-11-09 (Actual); Primary Completion 2017-05-31 (Actual); Study Completion 2017-07-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sairam Parthasarathy, MD, Principal Investigator — University of Arizona
Locations (1):
- University of Arizona School of Medicine, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A multi-site study that accrued over 2016 and into the middle of 2017.
Groups:
- Screening: All participants that consented to the study were considered for the participant flow. 15 participants were randomized to participate in the overnight in lab PSG's, these overnights were randomized to 1 of 4 interventions for each of the 4 overnights. This randomization scheme resulted in a large number of device sequences.
Period: Screening
Arm/Group | Screening
Started | 25
Completed | 15
Not Completed | 10
Not completed — Screen Failure | 10
Period: Overnight In-lab Polysomonography
Arm/Group | Screening
Started | 15
Modified Philips BiPAP ASV | 13
ResMed S7 VPAP Adapt | 13
Philips BiPAP AutoSV Advanced System One | 12
ResMed S9 VPAP Adapt | 12
Completed | 13
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Reason not given | 1
Period: Take Home Period
Arm/Group | Screening
Started | 13
Completed | 13
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Five participants screened failed prior to collecting demographic information.
Groups:
- Screening: All participants that consented to the study.
Arm/Group | Screening
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.3 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 20
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Average Apnea Hypopnea Index Among Different Polysomnography Devices.
Description: The Apnea Hypopnea Index is the number of the apneas and hypopneas during one hour of sleep. The average of these events over one night were compared during each overnight device use.
Time Frame: 4 nights
Population: 1 participant was excluded because he did not meet the criteria to receive ASV.
Measure: Mean (Standard Deviation); unit: events per hour
Groups:
- Philips BiPAP AutoSV Advanced System One: Philips Bilevel Postitive Airway Perssure (BiPAP) AutoSV Advanced System One: Auto SV Auto Servo Ventilation is a mode of positive airway pressure used to treat obstructive and complex central sleep apnea. This devices is FDA approved and will be set according to a predetermined setting.
- Modified Philips BiPAP ASV: Modified Philips BiPAP AutoServoventilation (ASV): This Modified BiPAP ASV will be set to a predetermined setting. This is the investigational device.
- ResMed S7 VPAP Adapt: ResMed S7 Variable Positive Airway Pressure (VPAP) Adapt: This device is FDA approved and will be set to predetermined setting.
Arm/Group | Philips BiPAP AutoSV Advanced System One | Modified Philips BiPAP ASV | ResMed S7 VPAP Adapt | ResMed S9 VPAP Adapt
Number analyzed (Participants) | 12 | 13 | 13 | 12
events per hour | 18.4 (23.0) | 25.4 (25) | 24.1 (25.4) | 19.2 (23.1)

ADVERSE EVENTS:
Time Frame: 40 days
Groups:
- Philips BiPAP AutoSV Advanced System One: The Bi-Level Positive Airway Pressure system will be used and will be configured with these settings.
  P max: 30 EPAP min: 4 EPAPmax: 15 PS min: 0 PS max: 15 BiFlex: 2 Rate: Auto
  Philips BiPAP AutoSV Advanced System One: Auto SV Auto Servo Ventilation is a mode of positive airway pressure used to treat obstructive and complex central sleep apnea. This devices is FDA approved and will be set according to a predetermined setting.
- ResMed S7 VPAP Adapt: This is an FDA approved device and the following settings will be administered:
  EEP: 4 PSmin: 3 PSMax: 16
  ResMed S7 VPAP Adapt: This device is FDA approved and will be set to predetermined setting.
- ResMed S9 VPAP Adapt: This is an FDA approved device and the following settings will be administered:
  EPAP min: 4 EPAPmax: 15 PS min: 0 PS max: 20 Max Ramp: Off
  ResMed S9 VPAP Adapt: This device is FDA approved and will be set to predetermined setting.
- Take Home - Modified Philips BiPAP ASV: After the overnight PSGs participants took home the Modified Philips BiPAP ASV for 30 days.
Arm/Group | Philips BiPAP AutoSV Advanced System One | Modified Philips BiPAP ASV | ResMed S7 VPAP Adapt | ResMed S9 VPAP Adapt | Take Home - Modified Philips BiPAP ASV
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/13 | 0/13 | 0/12 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/13 | 0/13 | 0/12 | 0/13
Other Adverse Events (participants affected / at risk) | 1/12 | 0/13 | 3/13 | 0/12 | 1/13
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Philips BiPAP AutoSV Advanced System One (N=12) | Modified Philips BiPAP ASV (N=13) | ResMed S7 VPAP Adapt (N=13) | ResMed S9 VPAP Adapt (N=12) | Take Home - Modified Philips BiPAP ASV (N=13)
EKG abnormalities (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Paroxysmal Supraventricular Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
seziure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
non-sustained ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0
Supraventricular Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-22): https://cdn.clinicaltrials.gov/large-docs/38/NCT02808338/Prot_SAP_000.pdf